CLINICAL TRIAL: NCT06585813
Title: Multiple Implant Placement with Simultaneous Soft Tissue Augmentation Using a Volume-stable Collagen Matrix Compared to Autogenous Connective Tissue Graft: a Clinical, Histological and Volumetric Pilot Study
Brief Title: Implants Placement with Simultaneous Soft Tissue Augmentation Using a Collagen Matrix Compared to Connective Tissue Graft: a Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: USJ -2023-62
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Soft Tissue Thickness Arround Implants
Keywords: collagen matrix; dental implant; subepithelial connective tissue graft; soft tissue augmentation
MeSH Terms: interventions — Dental Implants; Labor Stage, Second

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fibrogide group (Experimental): we are comparing the grafting of fibrogide(VCMX) with the connective tissue graft on multiple implant placement
  Interventions: Procedure: dental implant; Procedure: Fibrogide membrane; Procedure: second stage
- Connective Tissue graft Group (Experimental)
  Interventions: Procedure: dental implant; Procedure: connective tissue graft; Procedure: second stage

INTERVENTIONS:
Procedure: dental implant — we placed our implants and simultaneously grafted either fibroguide or CTG and after 3 months we did the second stage surgery
Procedure: Fibrogide membrane — we were comparing the efficacy of Fibrogide with the Connective tissue graft
  Arms: Fibrogide group
Procedure: connective tissue graft — the control group was the connective tissue graft group and the test group was the Fibrogide group
  Arms: Connective Tissue graft Group
Procedure: second stage — second stage to determine the thickness gained after the graft and to place a healing abutment

SUMMARY:
Background: To our knowledge, no study evaluated the use of VCMX at multiple implant sites and compared its efficacy and safety to a SCTG with the same dimensions. Therefore, we propose in the present protocol to evaluate the efficacy of VMCX to increase the thickness and height of soft tissue when placed at the time of multiple implant placement, as compared to SCTG.

Material and Methods: This study will be conducted in the saint joseph university periodontology department on at least 5 to 10 patients. The studied sites are the edentulous posterior mandible in a split-mouth model. The test groups are the groups grafted with VCMX and the control groups are the groups grafted with SCTG.

Some studies have been reported to compare these two techniques. But the specificity of our study is soft tissue augmentation on multiple implant sites in a split-mouth design.

ELIGIBILITY:
Inclusion Criteria:

* Adults ;18 years old.
* Patients with adequate oral hygiene (FMPI<20% and FMBI<20%).
* Healed implant sites (tooth extraction at least 8 to 12 weeks before enrolment).
* Patients who need prosthetic rehabilitation of at least two implants in the left and right posterior mandibular area.
* Inadequate amount of soft tissue where the implants are planned to be placed: thin mucosal tissues covering the edentulous alveolar ridge.
* Compliant patients are willing to sign an informed consent.

Exclusion Criteria:

* Uncontrolled periodontal disease.
* Heavy smoker (>10 cigarettes per day).
* General contraindications for dental surgical treatment.
* Insufficient bone volume for implant placement requiring bone augmentation procedures.
* History of malignancy, radiotherapy, or chemotherapy for malignancy within the past 5 years.
* Pregnancy or breastfeeding.
* Previous and concurrent medication affecting bone and mucosal healing.
* Disease affecting bone and connective tissue metabolism.
* Immediate implant placement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
keratinized tissue height | at the day of the surgery and after 3 months
  we will calculate the keratinized tissue height before the 1st surgery and before the 2nd stage with a periodontal probe
mucosal thickness | at the day of the surgery and after 3 months
  when doing the1st surgery(implant placement and soft tissue graft) and at the 2nd stage we will perform a mid crestal incision and reflect only the buccal flap , we will then with a periodontal probe calculate the peri-implant soft tissue thickness of the lingual flap (that we did not reflect). finally we will compare both measurments.

SECONDARY OUTCOMES:
time of the surgery | during the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nada Naaman, DDS,Msc in periodontology,PHD, Study Director — Saint-Joseph University /American University of Baghdad
Locations (1):
- Saint-Joseph University, Beirut, Beyrouth, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided